CLINICAL TRIAL: NCT00819663
Title: Intestinal Wall Remodeling After Initiation of Infliximab Therapy in Crohn's Disease Patients Undergoing Serial CT Enterography
Brief Title: Intestinal Wall Remodeling (Infliximab Therapy) in Crohn's Disease Patients Undergoing Serial Computed Tomography (CT) Enterography
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Centocor Ortho Biotech Services, L.L.C. (Industry)
Responsible Party: David H. Bruining, MD, Mayo Clinic Rochester, MN
Other Study IDs: 08-007338
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Crohns patients: Established Crohn's disease patients who underwent CTE imaging before and after initiating infliximab therapy

SUMMARY:
Anti-TNF therapy induces intestinal wall remodeling that correlates with clinical response and can be detected in patients undergoing serial computed tomography enterography (CTE).

DETAILED DESCRIPTION:
We will retrospectively identify Crohn's disease patients who underwent serial CTE imaging between 2004 and 2008. Approximately 4500 CTEs were performed over this period. We estimate a sample size of 50 Crohn's disease patients who have had CTE performed before and after infliximab therapy was initiated. We will analyze each CTE for the presence of penetrating disease, number of inflammatory lesion, length of each lesion, and severity of each lesion (degree of enhancement, wall thickness, stratification, vascular engorgement, fatty proliferation, and symmetry). Degree of enhancement and thickness will be graded on a 5-point scale. Stratification, vascular engorgement, fatty proliferation, and symmetry will be treated as dichotomous variables (yes/no). Only small bowel lesions will be described. A GI radiologist (JGF), blinded to the clinical information and previous imaging results, will provide the readings. Comparisons between CTEs will be performed to determine responders (all lesions improved), mixed responders (not all lesions improved), and refractory (no lesion improved). A descriptive pattern of healing will also be recorded for each lesion. Clinical data to be recorded include indication for CTE, time between CTE, dates of each CTE, date on first infliximab infusion, dose of infliximab, interval between infusions, history of penetrating disease, history of surgery, clinical status at imaging (remission, flare, or uncertain), medication usage, age, and disease duration. Clinical status at time of imaging will be based on the ordering clinician's global assessment at the time of repeat CTE. This will be determined by a review of the medical record by a gastroenterologist (DHB).

ELIGIBILITY:
Inclusion criteria

* Established Crohn's disease
* CTE before and after initiating infliximab
* Underwent at least 2 CTEs between 1/1/2004 and 12/31/2007
* At least 6 months between CTEs

  *off-label use of infliximab by either increased dose or shortened interval will be included in the study Exclusion criteria
* Small bowel surgery occurring before repeat CTE imaging
* Episodic infliximab therapy (intervals greater than every 8 weeks)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (Retrospectively) Established Crohn's disease patients who underwent CTE imaging before and after initiating infliximab therapy.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2009-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Anti-TNF therapy induces intestinal wall remodeling that correlates with clinical response and can be detected in patients undergoing serial computed tomography enterography (CTE). | 2004-2008

CONTACTS AND LOCATIONS:
Overall Officials: David H Bruining, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Bruining DH, Loftus EV Jr, Ehman EC, Siddiki HA, Nguyen DL, Fidler JL, Huprich JE, Mandrekar JN, Harmsen WS, Sandborn WJ, Fletcher JG. Computed tomography enterography detects intestinal wall changes and effects of treatment in patients with Crohn's disease. Clin Gastroenterol Hepatol. 2011 Aug;9(8):679-683.e1. doi: 10.1016/j.cgh.2011.04.025. Epub 2011 May 5. PMID 21621641